CLINICAL TRIAL: NCT04504032
Title: A Randomized, Controlled, Phase 2b Study to Evaluate Safety and Efficacy of Rivaroxaban (Xarelto®) for High Risk People With Mild COVID-19
Brief Title: A Trial to Evaluate Safety and Efficacy of Rivaroxaban (COVID-19)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on Data Monitoring Committee''s recommendation on 3 February 2021, the study was stopped on 4 February 2021 due to futility.
Sponsor: Gates Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gates MRI - COD-01-T01-01; 2020-005395-35 (EudraCT Number)
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: Rivaroxaban; Xarelto; Coronavirus; COVID-19; Coronavirus disease 2019
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental)
  Interventions: Drug: Rivaroxaban
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban — Participants self-administered rivaroxaban, 10 milligrams (mg) (1 tablet) orally once daily for 21 days.
  Arms: Rivaroxaban
Drug: Placebo — Participants self-administered rivaroxaban matching placebo orally once daily for 21 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess safety and clinical efficacy of rivaroxaban in people with mild Coronavirus Disease 2019 who are at increased risk of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at high-risk for Coronavirus disease 2019 (COVID-19) disease progression by fulfilling at least one of the following criteria at screening:

  * Presence of chronic pulmonary disease, chronic obstructive pulmonary disease (COPD), pulmonary hypertension
  * Diabetes mellitus (type 1 or type 2), requiring oral medication or insulin for treatment
  * Hypertension, requiring at least one oral medication for treatment
  * Immunocompromised status due to disease (e.g., those living with human immunodeficiency virus with a cluster of differentiation 4 [CD4] T-cell count of <200 per cubic millimeter [mm^3])
  * Immunocompromised status due to medication (e.g., taking 20 milligram [mg] or more of prednisone equivalents a day, anti-inflammatory monoclonal antibody therapies, cancer therapies)
  * Any chronic disease that is associated with high risk for severe COVID in the opinion of the site investigator
  * Body mass index ≥35 Kilogram per square meter (kg/m^2) (based on self-reported weight and height).
* Documented Severe Acute Respiratory Syndrome Coronavirus 2 positive diagnostic test of ≤7 days at the time of screening
* Symptomatic for COVID-19 for ≤72 hours at the time of screening (defined as having at least 2 of the following symptoms of COVID-19 that is of new onset or has worsened from baseline, and include fever, chills, myalgia, arthralgia, headache, fatigue, cough, sore throat, nasal congestion, anosmia, ageusia, nausea, vomiting, or diarrhea. If only two symptoms are present, they cannot both be anosmia and ageusia)
* Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the inform consent form and in this protocol
* Agree to participate in all remote, in-person or home visits as required in the protocol and provide updated contact information as necessary.
* Female of childbearing potential must agree to practice adequate contraception during the study

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Currently hospitalized or under immediate consideration for hospitalization at screening and Day 1
* Have new onset shortness of breath or increased shortness of breath from pre-COVID-19 (for people with known COPD) at screening and Day 1
* Hypoxemia (oxygen saturation <94% in ambient air or oxygen saturation below pre-COVID-19 level for people with known COPD) at Day 1
* Require supplemental oxygen (new requirement or increase in requirement from pre-COVID-19 condition) at screening and Day 1
* Have a history of (in the past 3 months) or current active pathological bleeding
* Have a history of hemorrhagic stroke or intracranial hemorrhage
* Have a recent severe head trauma within 30 days which includes concussion, skull fracture or hospitalization for head injury
* Have known intracranial neoplasm, cerebral metastases, arteriovenous malformation or aneurysm
* Have history of pregnancy-related hemorrhage
* Have active gastroduodenal ulcer or other gastrointestinal bleeding diagnosed in the past 3 months
* Currently are in a hemodynamically unstable state
* Currently require thrombolysis or pulmonary embolectomy
* Have history of severe hypersensitivity reaction to Xarelto®
* Currently have a prosthetic heart valve
* Have known diagnosis of triple positive antiphospholipid syndrome
* Have known diagnosis of chronic kidney disease (stage IV or receiving dialysis)
* Have a history of thrombocytopenia or known platelet count <100,000 cells/mm^3
* Have history of bronchiectasis and pulmonary cavitation
* Have active cancer (e.g, receiving chemotherapy or treatment for complication of the active cancer)
* Had epidural or neuraxial anesthesia or spinal puncture in the past 2 weeks and plan to undergo these procedures during the study
* Had surgery in the past 4 weeks or plan to undergo surgery during the study
* Currently is pregnant or plans to become pregnant
* Currently is breastfeeding
* Share household with an enrolled participant in this study
* Co-enrollment in any clinical trial that includes prohibited procedures (spinal puncture or surgery) or that includes treatments within the same drug class as rivaroxaban or treatments for which co-administration with rivaroxaban are prohibited. Note that any co-enrollment other than this requires approval by the Sponsor. For any co-enrolled study, the total volume of blood samples collected across the studies should not exceed 275 milliliters (mL) in 4 weeks.
* Currently using and plan to use the following medications during the study

  * Rivaroxaban or drugs in the same class
  * Dual anti-platelets therapy
  * Other anticoagulants
  * Combined Permeability glycoprotein (P-gp) and cytochrome P450 3A (CYP3A) inhibitors and inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GatesMRI, Study Director — Gates Medical Research Institute
Locations (20):
- United States (17):
  - Woodland Research Northwest LLC - ERG - PPDS, Rogers, Arkansas
  - Science 37, Inc, Los Angeles, California
  - Allergy and Asthma Medical Group and Research Center - CRN - PPDS, San Diego, California
  - Invesclinic, LLC, Fort Lauderdale, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - LCC Medical Research - Miami - BTC - PPDS, Miami, Florida
  - Adult Medicine of Lake County, Mt. Dora, Florida
  - Providea Health Partners LLC, Evergreen Park, Illinois
  - Clinical Research Institute, Inc - CRN - PPDS, Minneapolis, Minnesota
  - Encompass Care, North Las Vegas, Nevada
  - Riverside Medical Group - Circuit- PPDS, Secaucus, New Jersey
  - Elmhurst Hospital Center, Elmhurst, New York
  - Harlem Hospital Center, New York, New York
  - NYC Health + Hospitals/Lincoln, The Bronx, New York
  - Premier Family Physicians - Austin - Hunt - PPDS, Austin, Texas
  - Village Health Partners - Plano - Hunt - PPDS, Plano, Texas
  - South Texas Allergy and Asthma Medical Professionals, San Antonio, Texas
- United Kingdom (3):
  - Boundary House Medical Centre, Sale, Cheshire
  - St Mary's Hospital - PPDS, London, City of London
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 538 participants were screened of which only 497 were randomized to treatment.
Groups:
- Rivaroxaban: Participants self-administered rivaroxaban 10 milligrams (mg) (1 tablet) orally once daily for 21 days.
Period: Overall Study
Arm/Group | Rivaroxaban | Placebo
Started | 246 | 251
Completed | 210 | 223
Not Completed | 36 | 28
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 6 | 9
Not completed — Protocol Violation | 2 | 0
Not completed — Study terminated by sponsor | 1 | 2
Not completed — Withdrawal by Subject | 9 | 11
Not completed — Disease progression prior to dosing | 15 | 3
Not completed — Drug supply issues | 1 | 1
Not completed — Progressed to moderate/severe COVID-19 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Placebo | Total
Number analyzed (Participants) | 246 | 251 | 497
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (12.28) | 48.6 (12.14) | 49.2 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 159 | 299
  Male | 106 | 92 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 46 | 95
  Not Hispanic or Latino | 197 | 201 | 398
  Unknown or Not Reported | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 1 | 1
  Black or African American | 17 | 19 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 219 | 222 | 441
  Mixed race | 0 | 0 | 0
  Other | 7 | 7 | 14
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 and Grade 4 Adverse Events (AEs) Through Day 35
Description: An AE is any untoward medical occurrence that occurs in a participant. An AE can be any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with treatment, whether considered related to the product. AEs may include the onset of a new illness or undesirable medical condition or the exacerbation of pre-existing medical conditions. AE severity was graded as Grade 3 (Severe) and Grade 4 (Potentially Life-threatening) per the specific toxicity grading by the Division of Acquired Immunodeficiency Syndrome (DAIDS) AE Grading Table.
Time Frame: Up to Day 35
Population: Safety Population: all participants randomly assigned to study intervention, who received the study intervention. Participants were grouped according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 219 | 230
Participants | 6 | 13

2. Primary Outcome: Number of Participants With AEs Resulting in Study Intervention Discontinuation Through Day 35
Description: An AE is any untoward medical occurrence that occurs in a participant. An AE can be any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with treatment, whether considered related to the product. AEs may include the onset of new illness or undesirable medical condition or the exacerbation of pre-existing medical conditions.
Time Frame: Up to Day 35
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 219 | 230
Participants | 4 | 5

3. Primary Outcome: Number of Participants With Serious Adverse Events Through Day 35
Description: A serious AE is any untoward medical occurrence or effect, that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; is an important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require intervention to prevent one of the other outcomes.
Time Frame: Up to Day 35
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 219 | 230
Participants | 2 | 7

4. Primary Outcome: Number of Participants Who Progressed to Moderate or Severe Disease or Higher Based on the Gates MRI Ordinal Scale Through Day 28
Description: Participants who progressed to a moderate or severe disease category or higher (Bill & Melinda Gates Medical Research Institute [Gates MRI] ordinal scale ≥3) are reported. Gates MRI scale scores are assessed on a 7-point scale: 1=Asymptomatic/symptoms similar to pre-COVID-19 status; 2=Mild; 3=Moderate or severe; 4=Critically ill; 5=Critically ill with invasive mechanical ventilation or extrapulmonary complication; 6=Critically ill with Extra-Corporeal Membrane Oxygenation (ECMO); 7=Death.
Time Frame: Up to Day 28
Population: Intent-to-Treat (ITT) Population: All participants assigned to study intervention, who received the study intervention. Participants were grouped according to the study intervention to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Participants | 46 | 44

5. Secondary Outcome: Median Time to Disease Resolution Based on Symptoms Resolution Through Day 28
Description: Time to disease resolution is defined as the time from the first dose to the date of symptoms resolution (new-onset Coronavirus Disease 2019 [COVID-19] symptoms resolved, and pre-existing symptoms returned to Baseline) through Day 28. Baseline refers to health status prior to contracting new-onset COVID-19 symptoms. The 95% confidence interval (CI) for median and quartiles of time to disease resolution were calculated using the Kaplan Meier estimates.
Time Frame: Up to Day 28
Population: ITT Population. Only those participants with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 132 | 122
Days | 21.0 [19.0 to 23.0] | 23.0 [20.0 to 27.0]

6. Secondary Outcome: Median Time to Disease Resolution Based on Viral Clearance and Symptoms Resolution Through Day 28
Description: Time to disease resolution is defined as the time from the first dose to the date of both viral clearance (two consecutive negative diagnostic tests) and symptoms resolution (new-onset COVID-19 symptoms resolved, and pre-existing symptoms returned to Baseline) through Day 28. Baseline refers to health status prior to contracting new-onset COVID-19 symptoms. The 95% CI for median and quartiles of time to disease resolution were calculated using the Kaplan Meier estimates.
Time Frame: Up to Day 28
Population: ITT Population. Only those participants with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 125 | 115
Days | 23.0 [21.0 to 26.0] | 26.0 [22.0 to 28.0]

7. Secondary Outcome: Number of Participants Who Progressed to Moderate or Severe Disease or Higher Based on the Gates MRI Ordinal Scale at Day 8, 14, and 21
Description: Participants who progressed to a moderate or severe disease category or higher (Gates MRI ordinal scale ≥3) are reported. Gates MRI ordinal scale scores are assessed on a 7-point scale: 1=Asymptomatic/symptoms similar to pre-COVID-19 status; 2=Mild; 3=Moderate or severe; 4=Critically ill; 5=Critically ill with invasive mechanical ventilation or extrapulmonary complication; 6=Critically ill with ECMO; 7=Death.
Time Frame: Days 8, 14, and 21
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Participants
  Day 8 | 38 | 36
  Day 14 | 44 | 40
  Day 21 | 45 | 42

8. Secondary Outcome: Number of Participants Who Achieved Disease Resolution Based on Symptoms Resolution at Days 8, 14, 21, and 28
Description: Symptoms resolution is defined as new-onset COVID-19 symptoms resolved, and pre-existing symptoms returned to Baseline. Baseline refers to health status prior to contracting new-onset COVID-19 symptoms.
Time Frame: Days 8, 14, 21, and 28
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Participants
  Day 8 | 26 | 30
  Day 14 | 64 | 59
  Day 21 | 100 | 93
  Day 28 | 132 | 122

9. Secondary Outcome: Number of Participants Who Achieved Disease Resolution Based on Viral Clearance and Symptoms Resolution at Days 8, 14, 21, and 28
Description: Viral clearance is defined as two consecutive negative diagnostic tests. Symptoms resolution is defined as new-onset COVID-19 symptoms resolved, and pre-existing symptoms returned to Baseline. Baseline refers to health status prior to contracting new-onset COVID-19 symptoms.
Time Frame: Days 8, 14, 21, and 28
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Participants
  Day 8 | 12 | 20
  Day 14 | 49 | 44
  Day 21 | 86 | 83
  Day 28 | 125 | 115

10. Secondary Outcome: Number of Participants With the Indicated Gates Medical Research Institute (MRI) Scale Clinical Status at Days 8, 14, 21, and 28
Description: as for outcome 7
Time Frame: Days 8, 14, 21, and 28
Population: ITT Population. Only those participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Participants
  Day 8: number analyzed (Participants) | 188 | 198
  Day 8: Score 1 | 33 | 31
  Day 8: Score 2 | 152 | 159
  Day 8: Score 3 | 3 | 8
  Day 8: Score 4 | 0 | 0
  Day 8: Score 5 | 0 | 0
  Day 8: Score 6 | 0 | 0
  Day 8: Score 7 | 0 | 0
  Day 14: number analyzed (Participants) | 186 | 194
  Day 14: Score 1 | 69 | 55
  Day 14: Score 2 | 114 | 132
  Day 14: Score 3 | 3 | 7
  Day 14: Score 4 | 0 | 0
  Day 14: Score 5 | 0 | 0
  Day 14: Score 6 | 0 | 0
  Day 14: Score 7 | 0 | 0
  Day 21: number analyzed (Participants) | 186 | 193
  Day 21: Score 1 | 98 | 79
  Day 21: Score 2 | 87 | 109
  Day 21: Score 3 | 1 | 5
  Day 21: Score 4 | 0 | 0
  Day 21: Score 5 | 0 | 0
  Day 21: Score 6 | 0 | 0
  Day 21: Score 7 | 0 | 0
  Day 28: number analyzed (Participants) | 183 | 193
  Day 28: Score 1 | 125 | 108
  Day 28: Score 2 | 57 | 81
  Day 28: Score 3 | 1 | 4
  Day 28: Score 4 | 0 | 0
  Day 28: Score 5 | 0 | 0
  Day 28: Score 6 | 0 | 0
  Day 28: Score 7 | 0 | 0

11. Secondary Outcome: Number of Participants With the Indicated World Health Organization (WHO) Ordinal Scale Clinical Status at Days 8, 14, 21, and 28
Description: The WHO ordinal scale score is used to analyze the overall burden of disease and disease severity using an 11-point scale ranging from 0 to 10: 0=Uninfected; No viral ribonucleic acid (RNA) detected; 1=Asymptomatic; viral RNA detected; 2=Symptomatic; independent; 3=Symptomatic; assistance needed; 4=Hospitalized; no oxygen therapy (for isolation only); 5=Hospitalized; oxygen by mask or nasal prongs; 6=Hospitalized; oxygen by non-invasive ventilation (NIV) or high flow; 7=Intubation and mechanical ventilation, partial pressure of oxygen (pO2)/fraction of inspired oxygen (FiO2) ≥150 or oxygen saturation (SpO2)/FiO2 ≥200; 8=Mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or Vasopressors; 9=Mechanical ventilation pO2/FiO2 <150 and vasopressors, dialysis, or ECMO; 10=Dead.
Time Frame: Days 8, 14, 21, and 28
Population: ITT Population. Only those participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Participants
  Day 8: number analyzed (Participants) | 188 | 198
  Day 8: Score 0 | 19 | 19
  Day 8: Score 1 | 14 | 12
  Day 8: Score 2 | 154 | 166
  Day 8: Score 3 | 0 | 1
  Day 8: Score 4 | 1 | 0
  Day 8: Score 5 | 0 | 0
  Day 8: Score 6 | 0 | 0
  Day 8: Score 7 | 0 | 0
  Day 8: Score 8 | 0 | 0
  Day 8: Score 9 | 0 | 0
  Day 8: Score 10 | 0 | 0
  Day 14: number analyzed (Participants) | 186 | 194
  Day 14: Score 0 | 56 | 40
  Day 14: Score 1 | 15 | 16
  Day 14: Score 2 | 115 | 137
  Day 14: Score 3 | 0 | 1
  Day 14: Score 4 | 0 | 0
  Day 14: Score 5 | 0 | 0
  Day 14: Score 6 | 0 | 0
  Day 14: Score 7 | 0 | 0
  Day 14: Score 8 | 0 | 0
  Day 14: Score 9 | 0 | 0
  Day 14: Score 10 | 0 | 0
  Day 21: number analyzed (Participants) | 186 | 193
  Day 21: Score 0 | 87 | 72
  Day 21: Score 1 | 12 | 8
  Day 21: Score 2 | 87 | 112
  Day 21: Score 3 | 0 | 1
  Day 21: Score 4 | 0 | 0
  Day 21: Score 5 | 0 | 0
  Day 21: Score 6 | 0 | 0
  Day 21: Score 7 | 0 | 0
  Day 21: Score 8 | 0 | 0
  Day 21: Score 9 | 0 | 0
  Day 21: Score 10 | 0 | 0
  Day 28: number analyzed (Participants) | 183 | 193
  Day 28: Score 0 | 117 | 106
  Day 28: Score 1 | 9 | 4
  Day 28: Score 2 | 57 | 82
  Day 28: Score 3 | 0 | 1
  Day 28: Score 4 | 0 | 0
  Day 28: Score 5 | 0 | 0
  Day 28: Score 6 | 0 | 0
  Day 28: Score 7 | 0 | 0
  Day 28: Score 8 | 0 | 0
  Day 28: Score 9 | 0 | 0
  Day 28: Score 10 | 0 | 0

12. Secondary Outcome: Number of Participants With Hospitalization Through Days 8, 14, 21, and 28
Description: Participants who had clinical worsening and who had at least one hospitalization during the study were analyzed.
Time Frame: Days 8, 14, 21, and 28
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Participants
  Up to Day 8 | 3 | 6
  Up to Day 14 | 3 | 7
  Up to Day 21 | 3 | 7
  Up to Day 28 | 3 | 7

13. Secondary Outcome: Median Number of Days of Hospitalization Through Day 35
Description: Participants who had clinical worsening and who had at least one hospitalization during the study were analyzed. Hospitalized participants without an end date of hospitalization were not included.
Time Frame: Up to Day 35
Population: ITT Population
Measure: Median (Full Range); unit: Days
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Days | 5.0 [4.0 to 5.0] | 4.0 [2.0 to 30.0]

14. Secondary Outcome: Shift in Gates Medical Research Institute Ordinal Scale Score at Days 8, 14, 21, and 28
Description: Gates MRI ordinal scale scores are assessed on a 7-point scale: 1=Asymptomatic/symptoms similar to pre-COVID-19 status; 2=Mild; 3=Moderate or severe; 4=Critically ill; 5=Critically ill with invasive mechanical ventilation or extrapulmonary complication; 6=Critically ill with ECMO; 7=Death. BS= Baseline; PBS= Post-Baseline; NA= Data not available.
Time Frame: Days 8, 14, 21, and 28
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Participants
  Day 8: shift from BS score 1 to PBS score 1 | 2 | 1
  Day 8: shift from BS score 1 to PBS score 2 | 0 | 0
  Day 8: shift from BS score 1 to PBS score 3 | 0 | 0
  Day 8: shift from BS score 1 to PBS score >=4 | 0 | 0
  Day 8: shift from BS score 1 to PBS score NA | 0 | 0
  Day 8: shift from BS score 2 to PBS score 1 | 31 | 30
  Day 8: shift from BS score 2 to PBS score 2 | 152 | 158
  Day 8: shift from BS score 2 to PBS score 3 | 3 | 8
  Day 8: shift from BS score 2 to PBS score >=4 | 0 | 0
  Day 8: shift from BS score 2 to PBS score NA | 7 | 4
  Day 8: shift from BS score 3 to PBS score 1 | 0 | 0
  Day 8: shift from BS score 3 to PBS score 2 | 0 | 0
  Day 8: shift from BS score 3 to PBS score 3 | 0 | 0
  Day 8: shift from BS score 3 to PBS score >=4 | 0 | 0
  Day 8: shift from BS score 3 to PBS score NA | 12 | 3
  Day 8: shift from BS score NA to PBS score 1 | 0 | 0
  Day 8: shift from BS score NA to PBS score 2 | 0 | 0
  Day 8: shift from BS score NA to PBS score 3 | 0 | 0
  Day 8: shift from BS score NA to PBS score >=4 | 0 | 0
  Day 8: shift from BS score NA to PBS score NA | 15 | 17
  Day 14: shift from BS score 1 to PBS score 1 | 2 | 1
  Day 14: shift from BS score 1 to PBS score 2 | 0 | 0
  Day 14: shift from BS score 1 to PBS score 3 | 0 | 0
  Day 14: shift from BS score 1 to PBS score >=4 | 0 | 0
  Day 14: shift from BS score 1 to PBS score NA | 0 | 0
  Day 14: shift from BS score 2 to PBS score 1 | 67 | 54
  Day 14: shift from BS score 2 to PBS score 2 | 114 | 131
  Day 14: shift from BS score 2 to PBS score 3 | 3 | 7
  Day 14: shift from BS score 2 to PBS score >=4 | 0 | 0
  Day 14: shift from BS score 2 to PBS score NA | 9 | 8
  Day 14: shift from BS score 3 to PBS score 1 | 0 | 0
  Day 14: shift from BS score 3 to PBS score 2 | 0 | 1
  Day 14: shift from BS score 3 to PBS score 3 | 0 | 0
  Day 14: shift from BS score 3 to PBS score >=4 | 0 | 0
  Day 14: shift from BS score 3 to PBS score NA | 12 | 3
  Day 14: shift from BS score NA to PBS score 1 | 0 | 0
  Day 14: shift from BS score NA to PBS score 2 | 0 | 0
  Day 14: shift from BS score NA to PBS score 3 | 0 | 0
  Day 14: shift from BS score NA to PBS score >=4 | 0 | 0
  Day 14: shift from BS score NA to PBS score NA | 15 | 17
  Day 21: shift from BS score 1 to PBS score 1 | 2 | 0
  Day 21: shift from BS score 1 to PBS score 2 | 0 | 0
  Day 21: shift from BS score 1 to PBS score 3 | 0 | 0
  Day 21: shift from BS score 1 to PBS score >=4 | 0 | 0
  Day 21: shift from BS score 1 to PBS score NA | 0 | 1
  Day 21: shift from BS score 2 to PBS score 1 | 96 | 78
  Day 21: shift from BS score 2 to PBS score 2 | 87 | 109
  Day 21: shift from BS score 2 to PBS score 3 | 1 | 5
  Day 21: shift from BS score 2 to PBS score >=4 | 0 | 0
  Day 21: shift from BS score 2 to PBS score NA | 9 | 8
  Day 21: shift from BS score 3 to PBS score 1 | 0 | 1
  Day 21: shift from BS score 3 to PBS score 2 | 0 | 0
  Day 21: shift from BS score 3 to PBS score 3 | 0 | 0
  Day 21: shift from BS score 3 to PBS score >=4 | 0 | 0
  Day 21: shift from BS score 3 to PBS score NA | 12 | 3
  Day 21: shift from BS score NA to PBS score 1 | 0 | 0
  Day 21: shift from BS score NA to PBS score 2 | 0 | 0
  Day 21: shift from BS score NA to PBS score 3 | 0 | 0
  Day 21: shift from BS score NA to PBS score >=4 | 0 | 0
  Day 21: shift from BS score NA to PBS score NA | 15 | 17
  Day 28: shift from BS score 1 to PBS score 1 | 2 | 1
  Day 28: shift from BS score 1 to PBS score 2 | 0 | 0
  Day 28: shift from BS score 1 to PBS score 3 | 0 | 0
  Day 28: shift from BS score 1 to PBS score >=4 | 0 | 0
  Day 28: shift from BS score 1 to PBS score NA | 0 | 0
  Day 28: shift from BS score 2 to PBS score 1 | 123 | 106
  Day 28: shift from BS score 2 to PBS score 2 | 57 | 81
  Day 28: shift from BS score 2 to PBS score 3 | 1 | 4
  Day 28: shift from BS score 2 to PBS score >=4 | 0 | 0
  Day 28: shift from BS score 2 to PBS score NA | 12 | 9
  Day 28: shift from BS score 3 to PBS score 1 | 0 | 1
  Day 28: shift from BS score 3 to PBS score 2 | 0 | 0
  Day 28: shift from BS score 3 to PBS score 3 | 0 | 0
  Day 28: shift from BS score 3 to PBS score >=4 | 0 | 0
  Day 28: shift from BS score 3 to PBS score NA | 12 | 3
  Day 28: shift from BS score NA to PBS score 1 | 0 | 0
  Day 28: shift from BS score NA to PBS score 2 | 0 | 0
  Day 28: shift from BS score NA to PBS score 3 | 0 | 0
  Day 28: shift from BS score NA to PBS score >=4 | 0 | 0
  Day 28: shift from BS score NA to PBS score NA | 15 | 17

15. Secondary Outcome: Shift in World Health Organization Ordinal Scale Score at Days 8, 14, 21, and 28
Description: The WHO ordinal scale score is used to analyze the overall burden of disease and disease severity using an 11-point scale ranging from 0 to 10: 0=Uninfected; No viral ribonucleic acid (RNA) detected; 1=Asymptomatic; viral RNA detected; 2=Symptomatic; independent; 3=Symptomatic; assistance needed; 4=Hospitalized; no oxygen therapy (for isolation only); 5=Hospitalized; oxygen by mask or nasal prongs; 6=Hospitalized; oxygen by non-invasive ventilation (NIV) or high flow; 7=Intubation and mechanical ventilation, partial pressure of oxygen (pO2)/fraction of inspired oxygen (FiO2) ≥150 or oxygen saturation (SpO2)/FiO2 ≥200; 8=Mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or Vasopressors; 9=Mechanical ventilation pO2/FiO2 <150 and vasopressors, dialysis, or ECMO; 10=Dead. BS= Baseline; PBS= Post-Baseline; NA= Data not available.
Time Frame: Baseline; Days 8, 14, 21, and 28
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 222 | 222
Participants
  Day 8: shift from BS score 0 to PBS score 0 | 2 | 0
  Day 8: shift from BS score 0 to PBS score 1 | 0 | 0
  Day 8: shift from BS score 0 to PBS score 2 | 0 | 0
  Day 8: shift from BS score 0 to PBS score 3 | 0 | 0
  Day 8: shift from BS score 0 to PBS score 4 | 0 | 0
  Day 8: shift from BS score 0 to PBS score 5 | 0 | 0
  Day 8: shift from BS score 0 to PBS score >=6 | 0 | 0
  Day 8: shift from BS score 0 to PBS score NA | 0 | 0
  Day 8: shift from BS score 1 to PBS score 0 | 0 | 1
  Day 8: shift from BS score 1 to PBS score 1 | 0 | 0
  Day 8: shift from BS score 1 to PBS score 2 | 0 | 0
  Day 8: shift from BS score 1 to PBS score 3 | 0 | 0
  Day 8: shift from BS score 1 to PBS score 4 | 0 | 0
  Day 8: shift from BS score 1 to PBS score 5 | 0 | 0
  Day 8: shift from BS score 1 to PBS score >=6 | 0 | 0
  Day 8: shift from BS score 1 to PBS score NA | 0 | 0
  Day 8: shift from BS score 2 to PBS score 0 | 17 | 18
  Day 8: shift from BS score 2 to PBS score 1 | 14 | 12
  Day 8: shift from BS score 2 to PBS score 2 | 154 | 166
  Day 8: shift from BS score 2 to PBS score 3 | 0 | 1
  Day 8: shift from BS score 2 to PBS score 4 | 1 | 0
  Day 8: shift from BS score 2 to PBS score 5 | 0 | 0
  Day 8: shift from BS score 2 to PBS score >=6 | 0 | 0
  Day 8: shift from BS score 2 to PBS score NA | 18 | 7
  Day 8: shift from BS score 3 to PBS score 0 | 0 | 0
  Day 8: shift from BS score 3 to PBS score 1 | 0 | 0
  Day 8: shift from BS score 3 to PBS score 2 | 0 | 0
  Day 8: shift from BS score 3 to PBS score 3 | 0 | 0
  Day 8: shift from BS score 3 to PBS score 4 | 0 | 0
  Day 8: shift from BS score 3 to PBS score 5 | 0 | 0
  Day 8: shift from BS score 3 to PBS score >=6 | 0 | 0
  Day 8: shift from BS score 3 to PBS score NA | 1 | 0
  Day 8: shift from BS score NA to PBS score 0 | 0 | 0
  Day 8: shift from BS score NA to PBS score 1 | 0 | 0
  Day 8: shift from BS score NA to PBS score 2 | 0 | 0
  Day 8: shift from BS score NA to PBS score 3 | 0 | 0
  Day 8: shift from BS score NA to PBS score 4 | 0 | 0
  Day 8: shift from BS score NA to PBS score 5 | 0 | 0
  Day 8: shift from BS score NA to PBS score >=6 | 0 | 0
  Day 8: shift from BS score NA to PBS score NA | 15 | 17
  Day 14: shift from BS score 0 to PBS score 0 | 2 | 0
  Day 14: shift from BS score 0 to PBS score 1 | 0 | 0
  Day 14: shift from BS score 0 to PBS score 2 | 0 | 0
  Day 14: shift from BS score 0 to PBS score 3 | 0 | 0
  Day 14: shift from BS score 0 to PBS score 4 | 0 | 0
  Day 14: shift from BS score 0 to PBS score 5 | 0 | 0
  Day 14: shift from BS score 0 to PBS score >=6 | 0 | 0
  Day 14: shift from BS score 0 to PBS score NA | 0 | 0
  Day 14: shift from BS score 1 to PBS score 0 | 0 | 1
  Day 14: shift from BS score 1 to PBS score 1 | 0 | 0
  Day 14: shift from BS score 1 to PBS score 2 | 0 | 0
  Day 14: shift from BS score 1 to PBS score 3 | 0 | 0
  Day 14: shift from BS score 1 to PBS score 4 | 0 | 0
  Day 14: shift from BS score 1 to PBS score 5 | 0 | 0
  Day 14: shift from BS score 1 to PBS score >=6 | 0 | 0
  Day 14: shift from BS score 1 to PBS score NA | 0 | 0
  Day 14: shift from BS score 2 to PBS score 0 | 54 | 39
  Day 14: shift from BS score 2 to PBS score 1 | 15 | 16
  Day 14: shift from BS score 2 to PBS score 2 | 115 | 137
  Day 14: shift from BS score 2 to PBS score 3 | 0 | 1
  Day 14: shift from BS score 2 to PBS score 4 | 0 | 0
  Day 14: shift from BS score 2 to PBS score 5 | 0 | 0
  Day 14: shift from BS score 2 to PBS score >=6 | 0 | 0
  Day 14: shift from BS score 2 to PBS score NA | 20 | 11
  Day 14: shift from BS score 3 to PBS score 0 | 0 | 0
  Day 14: shift from BS score 3 to PBS score 1 | 0 | 0
  Day 14: shift from BS score 3 to PBS score 2 | 0 | 0
  Day 14: shift from BS score 3 to PBS score 3 | 0 | 0
  Day 14: shift from BS score 3 to PBS score 4 | 0 | 0
  Day 14: shift from BS score 3 to PBS score 5 | 0 | 0
  Day 14: shift from BS score 3 to PBS score >=6 | 0 | 0
  Day 14: shift from BS score 3 to PBS score NA | 1 | 0
  Day 14: shift from BS score NA to PBS score 0 | 0 | 0
  Day 14: shift from BS score NA to PBS score 1 | 0 | 0
  Day 14: shift from BS score NA to PBS score 2 | 0 | 0
  Day 14: shift from BS score NA to PBS score 3 | 0 | 0
  Day 14: shift from BS score NA to PBS score 4 | 0 | 0
  Day 14: shift from BS score NA to PBS score 5 | 0 | 0
  Day 14: shift from BS score NA to PBS score >=6 | 0 | 0
  Day 14: shift from BS score NA to PBS score NA | 15 | 17
  Day 21: shift from BS score 0 to PBS score 0 | 2 | 0
  Day 21: shift from BS score 0 to PBS score 1 | 0 | 0
  Day 21: shift from BS score 0 to PBS score 2 | 0 | 0
  Day 21: shift from BS score 0 to PBS score 3 | 0 | 0
  Day 21: shift from BS score 0 to PBS score 4 | 0 | 0
  Day 21: shift from BS score 0 to PBS score 5 | 0 | 0
  Day 21: shift from BS score 0 to PBS score >=6 | 0 | 0
  Day 21: shift from BS score 0 to PBS score NA | 0 | 0
  Day 21: shift from BS score 1 to PBS score 0 | 0 | 0
  Day 21: shift from BS score 1 to PBS score 1 | 0 | 0
  Day 21: shift from BS score 1 to PBS score 2 | 0 | 0
  Day 21: shift from BS score 1 to PBS score 3 | 0 | 0
  Day 21: shift from BS score 1 to PBS score 4 | 0 | 0
  Day 21: shift from BS score 1 to PBS score 5 | 0 | 0
  Day 21: shift from BS score 1 to PBS score >=6 | 0 | 0
  Day 21: shift from BS score 1 to PBS score NA | 0 | 1
  Day 21: shift from BS score 2 to PBS score 0 | 85 | 72
  Day 21: shift from BS score 2 to PBS score 1 | 12 | 8
  Day 21: shift from BS score 2 to PBS score 2 | 87 | 112
  Day 21: shift from BS score 2 to PBS score 3 | 0 | 1
  Day 21: shift from BS score 2 to PBS score 4 | 0 | 0
  Day 21: shift from BS score 2 to PBS score 5 | 0 | 0
  Day 21: shift from BS score 2 to PBS score >=6 | 0 | 0
  Day 21: shift from BS score 2 to PBS score NA | 20 | 11
  Day 21: shift from BS score 3 to PBS score 0 | 0 | 0
  Day 21: shift from BS score 3 to PBS score 1 | 0 | 0
  Day 21: shift from BS score 3 to PBS score 2 | 0 | 0
  Day 21: shift from BS score 3 to PBS score 3 | 0 | 0
  Day 21: shift from BS score 3 to PBS score 4 | 0 | 0
  Day 21: shift from BS score 3 to PBS score 5 | 0 | 0
  Day 21: shift from BS score 3 to PBS score >=6 | 0 | 0
  Day 21: shift from BS score 3 to PBS score NA | 1 | 0
  Day 21: shift from BS score NA to PBS score 0 | 0 | 0
  Day 21: shift from BS score NA to PBS score 1 | 0 | 0
  Day 21: shift from BS score NA to PBS score 2 | 0 | 0
  Day 21: shift from BS score NA to PBS score 3 | 0 | 0
  Day 21: shift from BS score NA to PBS score 4 | 0 | 0
  Day 21: shift from BS score NA to PBS score 5 | 0 | 0
  Day 21: shift from BS score NA to PBS score >=6 | 0 | 0
  Day 21: shift from BS score NA to PBS score NA | 15 | 17
  Day 28: shift from BS score 0 to PBS score 0 | 2 | 0
  Day 28: shift from BS score 0 to PBS score 1 | 0 | 0
  Day 28: shift from BS score 0 to PBS score 2 | 0 | 0
  Day 28: shift from BS score 0 to PBS score 3 | 0 | 0
  Day 28: shift from BS score 0 to PBS score 4 | 0 | 0
  Day 28: shift from BS score 0 to PBS score 5 | 0 | 0
  Day 28: shift from BS score 0 to PBS score >=6 | 0 | 0
  Day 28: shift from BS score 0 to PBS score NA | 0 | 0
  Day 28: shift from BS score 1 to PBS score 0 | 0 | 1
  Day 28: shift from BS score 1 to PBS score 1 | 0 | 0
  Day 28: shift from BS score 1 to PBS score 2 | 0 | 0
  Day 28: shift from BS score 1 to PBS score 3 | 0 | 0
  Day 28: shift from BS score 1 to PBS score 4 | 0 | 0
  Day 28: shift from BS score 1 to PBS score 5 | 0 | 0
  Day 28: shift from BS score 1 to PBS score >=6 | 0 | 0
  Day 28: shift from BS score 1 to PBS score NA | 0 | 0
  Day 28: shift from BS score 2 to PBS score 0 | 115 | 105
  Day 28: shift from BS score 2 to PBS score 1 | 9 | 4
  Day 28: shift from BS score 2 to PBS score 2 | 57 | 82
  Day 28: shift from BS score 2 to PBS score 3 | 0 | 1
  Day 28: shift from BS score 2 to PBS score 4 | 0 | 0
  Day 28: shift from BS score 2 to PBS score 5 | 0 | 0
  Day 28: shift from BS score 2 to PBS score >=6 | 0 | 0
  Day 28: shift from BS score 2 to PBS score NA | 23 | 12
  Day 28: shift from BS score 3 to PBS score 0 | 0 | 0
  Day 28: shift from BS score 3 to PBS score 1 | 0 | 0
  Day 28: shift from BS score 3 to PBS score 2 | 0 | 0
  Day 28: shift from BS score 3 to PBS score 3 | 0 | 0
  Day 28: shift from BS score 3 to PBS score 4 | 0 | 0
  Day 28: shift from BS score 3 to PBS score 5 | 0 | 0
  Day 28: shift from BS score 3 to PBS score >=6 | 0 | 0
  Day 28: shift from BS score 3 to PBS score NA | 1 | 0
  Day 28: shift from BS score NA to PBS score 0 | 0 | 0
  Day 28: shift from BS score NA to PBS score 1 | 0 | 0
  Day 28: shift from BS score NA to PBS score 2 | 0 | 0
  Day 28: shift from BS score NA to PBS score 3 | 0 | 0
  Day 28: shift from BS score NA to PBS score 4 | 0 | 0
  Day 28: shift from BS score NA to PBS score 5 | 0 | 0
  Day 28: shift from BS score NA to PBS score >=6 | 0 | 0
  Day 28: shift from BS score NA to PBS score NA | 15 | 17

16. Other Pre Specified Outcome: Change From Baseline in Gates Medical Research Institute Ordinal Scale Score at Days 8, 14, 21, and 28
Description: Gates MRI ordinal scale scores are assessed on a 7-point scale: 1=Asymptomatic/symptoms similar to pre- COVID-19 status; 2=Mild; 3=Moderate or severe; 4=Critically ill; 5=Critically ill with invasive mechanical ventilation or extrapulmonary complication; 6=Critically ill with ECMO; 7=Death. Instead of change from baseline, shift in scores from baseline was measured and have been presented in outcome measure 14.
Time Frame: Baseline; Days 8, 14, 21, and 28
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change From Baseline in World Health Organization Ordinal Scale Score at Days 8, 14, 21, and 28
Description: The WHO ordinal scale score is used to analyze the overall burden of disease and disease severity using an 11-point scale ranging from 0 to 10: 0=Uninfected; No viral ribonucleic acid (RNA) detected; 1=Asymptomatic; viral RNA detected; 2=Symptomatic; independent; 3=Symptomatic; assistance needed; 4=Hospitalized; no oxygen therapy (for isolation only); 5=Hospitalized; oxygen by mask or nasal prongs; 6=Hospitalized; oxygen by non-invasive ventilation (NIV) or high flow; 7=Intubation and mechanical ventilation, partial pressure of oxygen (pO2)/fraction of inspired oxygen (FiO2) ≥150 or oxygen saturation (SpO2)/FiO2 ≥200; 8=Mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or Vasopressors; 9=Mechanical ventilation pO2/FiO2 <150 and vasopressors, dialysis, or ECMO; 10=Dead. Instead of change from baseline, shift in scores from baseline was measured and have been presented in outcome measure 16.
Time Frame: Baseline; Days 8, 14, 21, and 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent up to 14 days after the last dose of study treatment (Day 35).
Description: Analysis was performed in the Safety Population, comprised of all participants randomly assigned to study intervention, who received the study intervention. Participants were grouped according to the study intervention they actually received.
Arm/Group | Rivaroxaban | Placebo
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/230
Serious Adverse Events (participants affected / at risk) | 2/219 | 7/230
Other Adverse Events (participants affected / at risk) | 12/219 | 11/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (N=219) | Placebo (N=230)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Acute kidney injury (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (N=219) | Placebo (N=230)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 0 (0)
COVID -19/COVID-19 pneumonia/pneumonia (Infections and infestations) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Hematuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Based on Data Monitoring Committee's recommendation on 3 February 2021, the study was stopped on 4 February 2021 due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT04504032/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT04504032/SAP_001.pdf